CLINICAL TRIAL: NCT02061228
Title: Endometrial Receptivity Enhancement Through Induced Injury and Repair During Ovarian Stimulation in an Antagonist Down-regulated Cycle
Brief Title: REFRESH: Receptivity Enhancement by Follicular-phase Renewal After Endometrial ScratcHing
Acronym: REFRESH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Safety concerns, apparent futility and protracted recruitment
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Samuel Santos-Ribeiro, MD, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 29012014REFRESH; 2014-000442-29 (EudraCT Number)
Record Dates: First submitted 2014-02-10; First posted 2014-02-12 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control arm (No Intervention): Women undergoing exogenous gonadotropin ovarian stimulation for ART in an antagonist downregulated cycle.
- Induced endometrial injury arm (Experimental): Women undergoing exogenous gonadotropin ovarian stimulation for ART in an antagonist downregulated cycle. Additionally, they will undergo an endometrial biopsy on the 6th day of ovarian stimulation using a Pipelle de Cornier® (CCD International, Paris, France).
  Interventions: Device: Pipelle de Cornier®

INTERVENTIONS:
Device: Pipelle de Cornier® — Women in the intervention group will undergo an endometrial biopsy on the 6th day of ovarian stimulation using a Pipelle de Cornier® (CCD International, Paris, France). This class I individually and sterile-packaged medical device, complies with Directive 93/42/European Economic Community (EEC) and is routinely used in our centre for endometrial sampling. It is comprised of a flexible disposable polypropylene suction cannula with an outer diameter of 3.1 mm and a 2.4 mm diameter opening on the distal end, on one side of the cannula. An inner plunger creates a vacuum essential for the blind endometrial biopsy. After the introduction of the Pipelle into the uterine cavity, it will be rotated 360 degrees and moved up and down four times after withdrawing the piston.
  Arms: Induced endometrial injury arm

SUMMARY:
A randomised controlled open-label clinical trial to assess the effect of artificially induced endometrial injury and repair during ovarian stimulation on the clinical pregnancy rate of an antagonist downregulated in-vitro fertilisation cycle

DETAILED DESCRIPTION:
Ovarian stimulation, ultrasound and hormonal monitoring, ovulation induction, oocyte retrieval, embryology procedure, IVF and luteal support will be according to how they are normally performed in our centre.

All women included will undergo artificial ovarian stimulation with gonadotropin-releasing hormone (GnRH) antagonist downregulation with daily injections of either ganirelix or cetrorelix. Treating physicians will opt on which exogenous gonadotropins should be used according to the patient's profile and preference and can include either recombinant follicle stimulating hormone (FSH) or highly purified urinary human menopausal gonadotropin (HP-HMG). Ovarian stimulation will commence after it is confirmed that the patient is not pregnant and has basal levels of oestradiol, progesterone, FSH and luteinizing hormone (LH). The stimulation will be monitored simultaneously by pelvic ultrasound and hormonal analysis (oestradiol, progesterone), starting on day 6 of stimulation and then every 1 to 3 days, according to the individual endocrine profile and follicular development.

Final oocyte maturation will be triggered with either 5000/10000 IU of human menopausal human chorionic gonadotropin (hCG) or 150 IU of recombinant hCG when more than 2 follicles of ≥17 mm are present. Oocyte retrieval will be performed 36 hours after hCG administration under either local anaesthesia with analgesic premedication or general anaesthesia, according to patient preference.

IVF or IVF/intracytoplasmatic sperm injection (ICSI) will be performed, using the specimen of sperm made available by the male progenitor on the day of oocyte retrieval. According to embryo quality, embryo transfer to the uterine cavity will be performed on either the 3rd or 5th day of development under ultrasound guidance whenever possible. Following embryo transfer, luteal support will be provided with vaginally administered progesterone 200 mg tid.

For clarity, cycle cancelation is defined as any interruption of the ART process that occurs before fresh embryo transfer. Cycle cancelation will occur a) upon patient request, b) if inadequate follicular development occurs, c) if no embryo is available for transfer.

ELIGIBILITY:
Inclusion Criteria:

* Fresh IVF/ICSI cycle
* Antagonist down-regulation
* Signed informed consent

Exclusion Criteria:

* Other known reasons for impaired implantation (i.e. hydrosalpinx, fibroid distorting the endometrial cavity, Asherman's syndrome, thrombophilia or endometrial tuberculosis)
* Oocyte donation acceptors
* Frozen egg transfers
* Embryos planned to undergo preimplantation genetic diagnosis (PGD)
* BMI >35 or <18
* Women already recruited for another trial on medically assisted procreation during the same cycle
* Women who have previously enrolled in the trial
* Those unable to comprehend the investigational nature of the proposed study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2014-03; Primary Completion 2018-02-26 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 12 weeks
  Sample size calculation was based on the adequate sample which would simultaneously 1) allow two safety-check interim analyses (at one-third and two-thirds of recruitment) and 2) have an 80% power to detect an increase of 15% in clinical pregnancy rate (from 32% to 47%) in the intervention group [using a two-side Fisher-exact test with a significance level (alfa) of 0.05]. Using a 1:1 randomisation ratio, each group would require approximately 180 patients, adding up to a total of 360 patients required for the trial.

SECONDARY OUTCOMES:
Live-birth rate | 42 weeks
  Delivery of at least one live born
Complication rate | 42 weeks
  Pain during biopsy, failed biospy and occurance of a premature delivery (<37 weeks) and low birth weight delivery (<2500 g)
Effect on the endometrial histology and expression | 2 weeks
  Histology and RNA expression analysis of collected samples

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Santos-Ribeiro, MD, Principal Investigator — Universitair Ziekenhuis Brussel; Shari Mackens, MD, Study Chair — Universitair Ziekenhuis Brussel; Dominic Stoop, PhD, Principal Investigator — Universitair Ziekenhuis Brussel; Herman Tournaye, PhD, Study Chair — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mackens S, Santos-Ribeiro S, Racca A, Daneels D, Koch A, Essahib W, Verpoest W, Bourgain C, Van Riet I, Tournaye H, Brosens JJ, Lee YH, Blockeel C, Van de Velde H. The proliferative phase endometrium in IVF/ICSI: an in-cycle molecular analysis predictive of the outcome following fresh embryo transfer. Hum Reprod. 2020 Jan 1;35(1):130-144. doi: 10.1093/humrep/dez218. PMID 31916571
- [Derived] Santos-Ribeiro S, Mackens S, Tournaye H, Blockeel C, Stoop D. Endometrial receptivity enhancement through induced injury and repair during ovarian stimulation: the Receptivity Enhancement by Follicular-phase Renewal after Endometrial ScratcHing (REFRESH) trial protocol. Hum Reprod Open. 2017 Nov 24;2017(3):hox022. doi: 10.1093/hropen/hox022. eCollection 2017. PMID 30895236